CLINICAL TRIAL: NCT03675360
Title: Low-Carbohydrate Dietary Pattern on Glycemic Outcomes Trial
Acronym: ADEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kirsten Dorans, Assistant Professor, Tulane University School of Public Health and Tropical Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-053; P20GM109036 (NIH)
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; PreDiabetes; Metabolic Disease; Hyperglycemia; Diet Modification; Glucose Intolerance; Glucose Metabolism Disorders (Including Diabetes Mellitus); Endocrine System Diseases
Keywords: Prediabetes; Diabetes; Low-Carbohydrate Diet
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Metabolic Diseases; Hyperglycemia; Glucose Intolerance; Glucose Metabolism Disorders; Endocrine System Diseases | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Carbohydrate Diet (Experimental): Behavioral modification to reduce carbohydrate consumption. Target <40 g net carbohydrates per day for first 3 months; <60 g net carbohydrates per day for months 4 onwards. The intervention will consist of 4 weekly individual counseling sessions, followed by 4 group sessions held every other week, with phone follow-ups in between group sessions. For the last 3 months of the study, there will be 3 monthly group sessions and 3 telephone follow-ups.
  At baseline, participants will receive written information with standard physical activity recommendations.
  Interventions: Behavioral: Low-Carbohydrate Diet
- Usual Diet (No Intervention): No dietary intervention.
  At baseline, participants will receive written information with standard dietary advice and standard physical activity recommendations.

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Behavioral modification to reduce carbohydrate consumption. Target <40 g net carbohydrates per day for first 3 months; <60 g net carbohydrates per day for months 4 onwards. The intervention will consist of 4 weekly individual counseling sessions, followed by 4 group sessions held every other week, with phone follow-ups in between group sessions. For the last 3 months of the study, there will be 3 monthly group sessions and 3 telephone follow-ups.
  At baseline, participants will receive written information with standard physical activity recommendations.
  Arms: Low-Carbohydrate Diet

SUMMARY:
The proposed randomized controlled trial will test the effect of a low-carbohydrate diet on hemoglobin A1c among individuals with elevated hemoglobin A1c that are within the range of prediabetes or diabetes. Results may provide evidence about the role of carbohydrate restriction in individuals with or at high risk of type 2 diabetes.

DETAILED DESCRIPTION:
In the short-term, among patients with type 2 diabetes, low-to-moderate carbohydrate diets have a greater glucose-lowering effect than do high-carbohydrate diets. However, compared with usual diet, the effect of a behavioral intervention promoting a low-carbohydrate/high-unsaturated fat and high-protein dietary pattern among individuals with prediabetes or untreated type 2 diabetes is not well understood.

The overall goal of this randomized controlled trial is to study the effect of a behavioral intervention promoting a low-carbohydrate/high-unsaturated fat and high-protein dietary pattern compared with usual diet on hemoglobin A1c (HbA1c) and other metabolic risk factors among individuals with or at high risk of diabetes (HbA1c 6.0-6.9%).

A total of 150 participants with HbA1c 6.0-6.9% will be recruited and randomly assigned to either a 6-month behavioral modification program designed to reduce carbohydrate intake (initial target <40 g digestible carbohydrates, final target <60 g digestible carbohydrates) or to usual diet in a 1:1 randomization ratio.

The primary outcome will be the difference between the active intervention and control groups for change in HbA1c from baseline to 6 months. Secondary outcomes will be fasting glucose, systolic blood pressure, total-to-high-density lipoprotein-cholesterol ratio, and body weight.

Findings from this study may provide evidence about the role of carbohydrate restriction in individuals with or at high risk of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 40 to 70 years
* HbA1c 6.0-6.9%
* Willing and able to provide informed consent

Exclusion Criteria:

* Diagnosed type 1 diabetes mellitus
* Use of agents affecting glycemic control (medications for diabetes, oral glucocorticoids) within the past three months prior to enrollment
* Medical condition in which low-carbohydrate diet may not be advised: estimated glomerular filtration rate (eGFR) ≤45 mL/min/1.73 m²; self-report of liver disease due to hepatitis or alcohol; osteoporosis; untreated thyroid disease; gout; cancer (other than non-melanoma skin cancer) requiring treatment in the past year, unless prognosis is excellent
* Factors that may affect HbA1c: hemoglobin <11 mg/dL (cutpoint for moderate-to-severe anemia, which could lead to falsely elevated or lowered HbA1c); recent blood donation or blood transfusion (self-report, past 4 months); human immunodeficiency virus (self-report)
* Self-reported history of intensive care unit stay due to Coronavirus Disease 2019 (COVID-19) in the past three months, as severe COVID-19 may affect blood glucose levels
* Allergies to nuts
* For women, current pregnancy, breastfeeding, or plans to become pregnant during the study
* Consumption of ≥21 alcoholic drinks per week or consumption of ≥6 drinks per occasion
* Current or planned residence making it difficult to meet trial requirements (due to distance from study site and/or challenges regularly traveling to site)
* Current participation in another lifestyle intervention trial or a pharmaceutical trial
* Participation of another household member in the study; employees or persons living with employees of the study
* Other concerns regarding ability to meet trial requirements, at the discretion of the principal investigator or study coordinator

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Dorans, ScD, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (1):
- Tulane Office of Health Research, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorans KS, Bazzano LA, Qi L, He H, Chen J, Appel LJ, Chen CS, Hsieh MH, Hu FB, Mills KT, Nguyen BT, O'Brien MJ, Samet JM, Uwaifo GI, He J. Effects of a Low-Carbohydrate Dietary Intervention on Hemoglobin A1c: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238645. doi: 10.1001/jamanetworkopen.2022.38645. PMID 36287562
- [Derived] Dorans KS, Bazzano LA, Qi L, He H, Appel LJ, Samet JM, Chen J, Mills KT, Nguyen BT, O'Brien MJ, Uwaifo GI, He J. Low-carbohydrate dietary pattern on glycemic outcomes trial (ADEPT) among individuals with elevated hemoglobin A1c: study protocol for a randomized controlled trial. Trials. 2021 Feb 1;22(1):108. doi: 10.1186/s13063-020-05001-x. PMID 33522954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from September 2018 through December 2020. Participants were recruited from the greater New Orleans, Louisiana area, primarily by mass mailing
Pre-assignment Details: After ascertaining eligibility, staff obtained randomization assignment in either a sealed envelope from or by telephoning the methodology unit at the time of randomization.
Groups:
- Low-Carbohydrate Diet: Behavioral modification to reduce carbohydrate consumption. Target <40 g net carbohydrates per day for first 3 months; <60 g net carbohydrates per day for months 4 onwards. The intervention will consist of 4 weekly individual counseling sessions, followed by 4 group sessions held every other week, with phone follow-ups in between group sessions. For the last 3 months of the study, there will be 3 monthly group sessions and 3 telephone follow-ups.
  At baseline, participants will receive written information with standard physical activity recommendations.
  Low-Carbohydrate Diet: Behavioral modification to reduce carbohydrate consumption. Target <40 g net carbohydrates per day for first 3 months; <60 g net carbohydrates per day for months 4 onwards. The intervention will consist of 4 weekly individual counseling sessions, followed by 4 group sessions held every other week, with phone follow-ups in between group sessions. For the last 3 months of the study, there will be 3 monthly group sessions and 3 telephone follow-ups.
  At baseline, participants will receive written information with standard physical activity recommendations.
Period: Overall Study
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Started | 75 | 75
Completed | 73 | 69
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Carbohydrate Diet | Usual Diet | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.0) | 58.6 (8.8) | 58.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 68 | 71 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 49 | 85
  White | 33 | 24 | 57
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
Body weight [Mean (Standard Deviation); unit: kg] | 102.6 (21.8) | 96.4 (19.6) | 99.5 (20.9)
Waist circumference [Mean (Standard Deviation); unit: cm] | 115.9 (14.8) | 111.8 (15.0) | 113.9 (15.0)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 6.17 (0.31) | 6.14 (0.30) | 6.16 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c
Description: 6-month change in Hemoglobin A1c comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Data were analyzed using intention to treat. For the primary outcome (net 6-month change in HbA1c), we used linear mixed effects models with HbA1c as the dependent variable. This model included a random intercept with an unstructured covariance matrix, indicator variables for time and study group, and group by time interaction terms.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
percentage | -0.26 [-0.33 to -0.19] | -0.04 [-0.10 to 0.02]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.32 to -0.14]

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: 6-month change in fasting plasma glucose comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat analysis.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
mg/dL | -8.4 [-12.3 to -4.4] | 1.9 [-1.8 to 5.5]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -10.3, 95% CI 2-sided [-15.6 to -4.9]

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: 6-month change in systolic blood pressure comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
mm Hg | -4.9 [-7.9 to -1.8] | -1.6 [-4.4 to 1.2]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -3.2, 95% CI 2-sided [-7.3 to 0.9]

4. Secondary Outcome: Change in Total-to-HDL-cholesterol Ratio
Description: 6-month change in total-to-HDL-cholesterol ratio comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
ratio | -0.54 [-0.67 to -0.40] | -0.41 [-0.52 to -0.29]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Median Difference (Final Values) = -0.13, 95% CI 2-sided [-0.31 to 0.05]

5. Secondary Outcome: Change in Body Weight
Description: 6-month change in body weight comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
kg | -6.4 [-7.8 to -5.1] | -0.5 [-1.2 to 0.2]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -5.9, 95% CI 2-sided [-7.4 to -4.4]

6. Other Pre Specified Outcome: Change in Insulin
Description: 6-month change in fasting insulin comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: μIU/L
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
μIU/L | -4.0 [-7.2 to -0.8] | 2.3 [-0.5 to 5.0]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -6.2, 95% CI 2-sided [-10.5 to -2.0]

7. Other Pre Specified Outcome: Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: 6-month change in HOMA-IR comparing low-carbohydrate arm with usual diet arm. HOMA-IR was calculated as fasting insulin (μIU/mL) x fasting glucose (mmol/L)/22.5.
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: no units
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
no units | -1.6 [-2.6 to -0.7] | 0.8 [-0.2 to 1.7]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -2.4, 95% CI 2-sided [-3.7 to -1.1]

8. Other Pre Specified Outcome: Change in Diastolic Blood Pressure
Description: 6-month change in diastolic blood pressure comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
mm Hg | -3.2 [-5.2 to -1.2] | -0.6 [-2.3 to 1.1]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -2.6, 95% CI 2-sided [-5.2 to 0]

9. Other Pre Specified Outcome: Change in Waist Circumference
Description: 6-month change in waist circumference comparing low-carbohydrate arm with usual diet arm
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
cm | -5.2 [-6.9 to -3.5] | -0.5 [-1.6 to 0.5]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -4.7, 95% CI 2-sided [-6.7 to -2.6]

10. Other Pre Specified Outcome: Change in Estimated Atherosclerotic Cardiovascular Disease Risk
Description: 6-month change in estimated 10-year atherosclerotic cardiovascular disease risk comparing low-carbohydrate arm with usual diet arm.
  The estimated 10-year cardiovascular disease risk was assessed by 2013 American College of Cardiology/American Heart Association Atherosclerotic Cardiovascular Disease Risk Score, known as the Pooled Cohort Equations. The Pooled Cohort Equations estimate the 10-year primary risk of ASCVD (atherosclerotic cardiovascular disease) among patients without pre-existing cardiovascular disease who are between 40 and 79 years of age. Variables included in the risk score include: gender, age, race, total cholesterol, HDL cholesterol, systolic blood pressure, treatment for blood pressure, diabetes, and smoking status.
  Reference: Goff DC, Lloyd-Jones DM et al. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: A report of the American college of cardiology/American heart association task force on practice guidelines. Vol. 129, Circulation. 2014.
Time Frame: Baseline and six months
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: estimated %
Arm/Group | Low-Carbohydrate Diet | Usual Diet
Number analyzed (Participants) | 75 | 75
estimated % | -1.7 [-2.5 to -0.9] | -0.9 [-1.6 to -0.2]
Statistical Analysis 1: Comparison: Low-Carbohydrate Diet vs Usual Diet; Test type: Superiority; p < 0.05, linear mixed effects model; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.8 to 0.3]

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was collected over the 6-month intervention period.
Arm/Group | Low-Carbohydrate Diet | Usual Diet
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 4/75 | 3/75
Other Adverse Events (participants affected / at risk) | 2/75 | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Carbohydrate Diet (N=75) | Usual Diet (N=75)
Emergency room visit (Infections and infestations) | 1 (1) | 1 (1)
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)
Emergency Room Visit (Vascular disorders) | 0 (0) | 1 (1)
Surgery and hospitalization (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Carbohydrate Diet (N=75) | Usual Diet (N=75)
Surgery (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Surgery (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03675360/Prot_SAP_000.pdf